CLINICAL TRIAL: NCT00822510
Title: Telephone Counseling With Men With Prostate Cancer and Partners
Brief Title: Telephone Counseling: Men With Prostate Cancer & Partners
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Terry Badger, Professor, University of Arizona
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04-0376-02; R21CA113409 (NIH)
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: Psychosocial Intervention; Men with Prostate Cancer & Partners
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone Interpersonal Counseling (Experimental): Telephone delivered interpersonal counseling support intervention. Intervention was for 8 weeks. Participants were called on the telephone each week for about 30 minutes.
  Interventions: Behavioral: Telephone Interpersonal Counseling
- Telephone delivered education only (Active Comparator): Telephone delivered education only. Educational topics included prostate cancer health, side effects, physical activity, diet. Participants were called on the telephone each week for about 30 minutes.
  Interventions: Behavioral: Telephone delivered education only

INTERVENTIONS:
Behavioral: Telephone Interpersonal Counseling — Telephone delivered 8 week education and counseling intervention based on interpersonal psychotherapy.
  Arms: Telephone Interpersonal Counseling
Behavioral: Telephone delivered education only — Telephone delivered 8 week educational intervention on prostate cancer health, side effects, physical activity, diet, smoking cessation
  Arms: Telephone delivered education only

SUMMARY:
The purpose of this project is to test a telephone delivered educational support program versus an education only program for improving symptom management and quality of life in men with prostate cancer and their partners.

DETAILED DESCRIPTION:
Eligibility Criteria for men: receiving treatment for prostate cancer,over 21 years of age, English speaking, have access to and ability to talk on the phone and have a partner willing to participate in the study. Participants can live anywhere in the United States because the intervention is telephone delivered.

Partners can be anyone the man selects (friend or relative) who is over 21 years of age, English speaking and has access to or ability to speak on the phone.

Men and their partners will be assigned to one of two groups. Each survivor will receive 8 telephone calls over an 8-week period for about 30 minutes each. Each partner will receive 4 telephone calls every other week for about 30 minutes each. We will ask everyone to complete a baseline assessment over the telephone, after the 8 weeks, and then again about 8 weeks after the second assessment.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment for prostate cancer
* Over 21 years
* Access to and ability to talk on the phone
* Speaks English and has a partner to participate with him.
* Partners are anyone who the man chooses (friend or relative) who is over 21 years, English speaking and has access and ability to talk on the phone.

Exclusion Criteria:

* under 21 years
* Does not speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Badger, PhD, RN, Principal Investigator — University of Arizona College of Nursing
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: College of Nursing Webpage — http://nursing.arizona.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone Delivered Interpersonal Counseling: Telephone delivered education and support for 8 weeks
  Telephone Interpersonal Counselling Intervention: Telephone delivered 8 week education and support intervention
- Telephone Delivered Education Only: Telephone delivered education only for 8 weeks
  Telephone delivered education only: Telephone delivered education for 8 weeks
Period: Overall Study
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Started | 38 | 41
Completed | 35 | 36
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.5) | 68.3 (9.6) | 66.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were asked if they were male or female
  Participants
    Female | 0 | 0 | 0
    Male | 38 | 41 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 35 | 38 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiological Studies-Depression Scale
Description: Depression was measured by the 20-item Center for Epidemiological Studies-Depression (CES-D) scale, Range is 0-60. Scores are added together with higher score greater depression.
Time Frame: 3 points in time, baseline, T2=T1+8 weeks, T3=T2 plus 8 weeks
Population: Badger, T.A., Segrin, C., Figueredo, A.J., Harrington, J., Sheppard, K., Passalacqua, S., Pasvogel, A., & Bishop, M. (2011) Psychosocial Interventions to Improve Quality of Life in Prostate Cancer Survivors and their Intimate or Family Partners. Quality of Life Research. 20 (6), 833-844 [epub Dec 2010]. PMID: 21170682; PMCID: PMC3117079
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 35 | 36
units on scale
  Time 1 | 11.41 (9.0) | 12.43 (9.7)
  Time 2 | 11.39 (9.2) | 9.06 (9.7)
  Time 3 | 11.18 (13.4) | 8.86 (10)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p < .05, ANOVA

2. Primary Outcome: Perceived Stress
Description: Perceived stress scale is a 10-item scale with a range of 0-40. Higher scores indicate more stress.
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 12.69 (6.5) | 13.17 (9.7)
  Time 2 | 12.45 (6.5) | 11.23 (7.3)
  Time 3 | 12.25 (7.1) | 9.9 (6.7)

3. Primary Outcome: Positive Affect
Description: Positive and Negative Affect Scale is a 20 item scale that measures positive and negative affect subscales. Scores range from 10-50 on each subscale with higher score indicating more positive affect.
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 35.11 (6.6) | 36.71 (7.4)
  Time 2 | 36.7 (7.7) | 37.87 (6.1)
  Time 3 | 35.84 (8.5) | 37.52 (6.7)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p = .79, ANOVA

4. Primary Outcome: Negative Affect
Description: as for outcome 3
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 15.97 (6.3) | 17.03 (7.4)
  Time 2 | 16.76 (7.1) | 14.84 (6.2)
  Time 3 | 15.32 (6.4) | 14.07 (4.1)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p = .001, ANOVA

5. Primary Outcome: Multidimensional Fatigue Inventory
Description: Measure of physical well-being, specifically fatigue, using the Multidimensional Fatigue Scale. Scores range from 0-80 with higher scores indicative of more fatigue.
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 26.78 (15.8) | 28.17 (18.1)
  Time 2 | 27.06 (17.5) | 24.48 (19.2)
  Time 3 | 26.81 (17.5) | 21.69 (17.5)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p = .001, ANOVA

6. Primary Outcome: Social Well Being
Description: Measures social well-being using the 9 item Social Well-being scale, ranging from 9-90. Higher score indicates increased social well-being.
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 56.31 (17.3) | 61.13 (16.1)
  Time 2 | 59.15 (15.7) | 62.71 (16.1)
  Time 3 | 56.66 (19.5) | 63.1 (16)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p = .71, ANOVA

7. Primary Outcome: Spiritual Well Being
Description: Measures if spiritual beliefs using a 7-item scale that ranges from 7-70. Higher score equals greater spiritual wellbeing.
Time Frame: 3 points in time, baseline, second assess (T1-8week), 3rd assessment (T2+8 weeks)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Number analyzed (Participants) | 36 | 34
units on scale
  Time 1 | 43.64 (14.8) | 44.17 (11.6)
  Time 2 | 42.76 (14) | 46.45 (11.9)
  Time 3 | 42.09 (13.9) | 47.83 (12)
Statistical Analysis 1: Comparison: Telephone Delivered Interpersonal Counseling vs Telephone Delivered Education Only; Test type: Superiority or Other; p = .01, ANOVA

ADVERSE EVENTS:
Time Frame: There were no adverse advents to report
Arm/Group | Telephone Delivered Interpersonal Counseling | Telephone Delivered Education Only
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No